CLINICAL TRIAL: NCT02729948
Title: Use of a Tethered Capsule Endoscope in Screening for Barrett's Esophagus
Brief Title: Tethered Capsule Endoscope in Screening Patients With Barrett Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 9561; NCI-2016-00112 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9561 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2016-03-25; First posted 2016-04-06 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Endoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Screening (TCE) (Experimental): Patients swallow the TCE and undergo endoscopic examination while they are seated on a standard endoscopy gurney. Patients undergo standard of care EGD on the same day.
  Interventions: Other: Survey Administration; Device: Tethered Capsule Endoscope

INTERVENTIONS:
Other: Survey Administration — Ancillary studies
Device: Tethered Capsule Endoscope — Undergo TCE
  Other Names: TCE

SUMMARY:
This pilot clinical trial studies how well tethered capsule endoscope works in screening patients with Barrett esophagus (BE), a condition where the lining of the esophagus has changed or has been replaced with abnormal cells that may lead to cancer also called esophageal cancer. In an attempt to prevent the progression from BE to esophageal cancer, patients undergo a standard procedure called esophagogastroduodenoscopy (EGD) where patients are sedated and the doctor uses an endoscope to examine the tissue in the esophagus. Tethered capsule endoscope is a tiny capsule with a laser scan inside and a very thin cord attached to it. Patients swallow the capsule and the thin cord keeps the capsule in specific area in the esophagus. After pictures of the lining of esophagus are taken, the capsule is removed using the thin cord. Tethered capsule endoscope may be able to identify tissue changes in patients with BE without the need for sedation or anesthesia, thus eliminating the associated risks and costs associated with EGD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate image quality and usability of the tethered capsule endoscope after repeated clinical use and reprocessing.

II. Evaluate safety issues associated with the use of the device for this subject population - was there any noticeable difference from prior study of subjects at high risk of Barrett's esophagus using the same device, but without reprocessing.

SECONDARY OBJECTIVES;

I. Study other specified device characteristics or device application considerations.

II. Obtain preliminary data for use in designing a subsequent pivotal study of the device.

OUTLINE:

Patients swallow the tethered capsule endoscope (TCE) and undergo endoscopic examination while they are seated on a standard endoscopy gurney. Patients undergo standard of care EGD on the same day.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent
* Scheduled for endoscopic screening and/or evaluation of Barrett's esophagus

Exclusion Criteria:

* Previous history of a swallowing disorder, such as scleroderma, achalasia, esophageal stricture or esophageal diverticulum
* Symptoms of dysphagia
* Suspicion or known history of gastrointestinal obstruction
* History of prior surgery on the oropharynx, neck, esophagus, or stomach
* Current diagnosis of cancer, unstable cardiovascular disease, end-stage liver or kidney disease, or other major medical illness
* Currently taking anticoagulant medications or clopidogrel
* Major physical disability which would prevent subject from transferring from a chair to a bed and sitting in an upright position
* Inability to abstain from taking anything by mouth for at least 6 hours
* Currently pregnant
* Expected to undergo magnetic resonance imaging (MRI) within two weeks following the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Consistent image quality | At the conclusion of TCE exam (day 1)
  Consistent image quality defined as no significant degradation of lateral spatial resolution [line pairs per mm] and axial depth of focus [mm], maximum field of view [degrees cone angle], and color fidelity [qualitatively matches color chart] when measured after use in the clinic using color and resolution test targets and a test chamber to measure field of view. The standard care EGD will be digitally recorded to allow for review and comparison to the TCE procedure by a blinded, expert endoscopist.
Consistent usability defined as no significant change to the tolerance rating given by the patient by survey, and ease of use by the physician by survey, and time for completing the examination | At the conclusion of TCE exam (day 1)
Incidence of adverse events associated with TCE use | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saunders, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States